CLINICAL TRIAL: NCT00299195
Title: A Pilot Multi-Center International Double-Blind Placebo Controlled Randomized Study of Sulindac, a Pan-Cox Inhibitor, in Oral Premalignant Lesions
Brief Title: A Randomized Study of Sulindac in Oral Premalignant Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: AIMS Institute (Other); Weill Medical College of Cornell University (Other); Regional Cancer Centre, Trivandrum, India (Other); Narayana Hrudayalaya Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-099
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-01

CONDITIONS: Leukoplakia, Oral; Benign Neoplasms
Keywords: Oral Leukoplakia; Benign Neoplasms; Chemoprevention; Pan-cyclooxygenase (COX) inhibitor; sulindac; 04-099
MeSH Terms: conditions — Leukoplakia, Oral; Neoplasms; Coproporphyria | interventions — Sulindac

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): sulindac
  Interventions: Drug: sulindac
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sulindac — Sulindac 150 mg po bid x 24 weeks
  Arms: 1
Drug: Placebo — Placebo bid x 24 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to see if a drug called sulindac can prevent the development of changes in the mouth that are related to oral pre-cancer growths (oral epithelial dysplasia) or oral cancer. Sulindac is an anti-inflammatory drug that has already been tested in people with arthritis (inflammation of a joint).

This study is being done by Memorial Sloan-Kettering Cancer Center in New York, Amrita Institute of Medical Sciences and Research Center in Cochin, India, and Regional Cancer Centre (RCC) in Trivandrum, India.

DETAILED DESCRIPTION:
Oral precancerous lesions (OPL) represent a valuable model for clinical trials for tobacco related cancers. However, due to the relatively low prevalence of this condition in the United States, subject accrual to such trials is slow. Conversely, in India, the prevalence of oral leukoplakia is among the highest in the world. Indeed oral cancer, caused by exposure to tobacco smoke, alcohol and betel nut quid, is the leading cause of cancer deaths in India.

To date, there are no effective treatments documented in randomized controlled clinical trials to prevent malignant transformation of leukoplakia. However, evidence that non-steroidal anti-inflammatory drugs (NSAIDs) prevent experimental and animal head and neck cancer, and colon and breast cancer in humans lends support to the promise of NSAIDs in the chemoprevention of oral cancer.

The purpose of this protocol is to pilot a multi-center chemoprevention trial of sulindac, a pan-cyclooxygenase (COX) inhibitor, for oral leukoplakia through an international collaboration between Memorial Sloan-Kettering Cancer Center (MSKCC), New York, Regional Cancer Centre (RCC) in Trivandrum, India and the Amrita Institute of Medical Sciences (AIMS), Kerala, India. Specifically, we will conduct a 66 subject, 2-arm, double-blind, placebo-controlled randomized study of sulindac 150 mg bid to test the clinical efficacy, safety and molecular effects of sulindac against OPL and OPL tissue. Oral leukoplakia subjects will be enrolled from both RCC, AIMS and MSKCC, however, we expect that most subjects will be recruited from AIMS due to the substantially higher prevalence of this condition among the Indian compared to the US population.

MSKCC will be the coordinating center for this trial, and will thus be responsible for all aspects of clinical trial design and management. Our study team, in collaboration with the Office of Clinical Research and the Office of the Physician-in-Chief, has spent a considerable amount of time and effort in developing a comprehensive data and safety monitoring (DSM) plan.

ELIGIBILITY:
Inclusion Criteria:

For this study an Oral Premalignant Lesions (OPL) is defined as a lesion which can include atypical hyperplasia, atypical hyperkeratosis, leukoplakia, and erythroplakia/erythro-leukoplakia. Histology MUST be confirmed by an MSKCC pathologist for all participating sites. An OPL may be located in the oral cavity, oropharynx.

* The subj has a histologically suspected or confirmed index oral premalignant lesion, 12mm or greater in size that has not been bx'd in the past 6 wks. Each index lesion must be either:

  * An EARLY premalignant lesion defined to be at high risk as indicated by the presence of at least one of the following: atypical cells or mild dysplasia, or hyperplastic leukoplakia of high-risk sites, lateral and ventral tongue and floor or mouth OR
  * An ADVANCED premalignant lesion defined as the presence of at least one of the following: moderate dysplasia or severe dysplasia (excluding CIS)
* The subj is > 18 yrs of age
* The subj's life expectancy is > 12 wks and Zubrod performance status is 0 or 1 (Appendix VIII).
* The subj meets the following lab eligibility criteria during a time not to exceed 4 wks prior to randomization.

  * Hemoglobin level above 10g/dL for women and above 12g/dL for men.
  * WBC count > 3,000 uL.
  * Platelets count > 125,000 uL.
  * Total bilirubin < or = 1.5xULN
  * AST (SGOT) and ALT (SGPT) < or = 2.5 x ULN.
  * BUN and serum creatinine < or = 1.5 x ULN.
* If the subj is female and of childbearing potential (women are considered not of childbearing potential if they are at least 2 yrs postmenopausal and/or surgically sterile), she:

  * has been using adequate contraception (abstinence, IUD, birth control pills, or spermicidal gel with diaphragm or condom) since her last menses and will use adequate contraception during the study, AND
  * is not lactating, AND
  * has a documented negative serum pregnancy test within 14 ds prior to randomization.
* The subj's history/use of NSAIDs, aspirin, corticosteroids meets the following criteria:

  * total oral/intravenous corticosteroid use has been < 14 ds within 6 mos of the Baseline visit, and
  * total inhaled corticosteroid use has been < 30 ds within 6 mos of the Baseline visit, and
  * is willing to limit aspirin use to < or = 120 mg po per d (typical cardioprotective dose in India) or < or = 80 mg po per d (typical cardioprotective dose in the US) for the duration of the study, and is willing to abstain from chronic use of all NSAIDs and COX-2 inhibitors for duration of study. Chronic use of NSAIDs is defined as a frequency of > or = 3 times/wk AND for more than a total of 14 ds a yr.
* The subj has discontinued any other chemopreventive therapy at least 3 mos prior to the Baseline visit and all toxicities have been fully resolved.
* If applicable, the subj has been counseled on smoking cessation.
* If the subject is male, will use adequate contraception during the study.

Exclusion Criteria:

* The subject has had chemotherapy, immunotherapy, hormonal tx (other than HRT for menopause), or RT within 3 wks of the Baseline visit.
* The subj has not recovered from the acute toxic effects of chemotherapy, immunotherapy, hormonal tx, or RT.
* The subj will need concurrent chemotherapy, radiotherapy, hormonal (other than HRT for menopause), or immunotherapy during the time of study.
* The subj has a history of hypersensitivity to sulindac, COX-2 inhibitors, NSAIDs, salicylates.
* The subj has been diagnosed with or has been treated for esophageal, gastric, pyloric channel, or duodenal ulceration.
* The subj has a history of inv cancer within the past 1 yr (excluding non-melanoma skin cancer and in situ cervical cancer).
* The subj has a chronic or acute renal or hepatic disorder or a significant bleeding disorder or any other condition which, in the Institutional Principal Investigator's opinion, might preclude study participation.
* The subj has a past history of or active inflammatory bowel disease (eg. Crohn's disease or ulcerative colitis) or pancreatic disease.
* The subj has received any investigational medication within 30 ds of the Baseline visit or is scheduled to receive an investigational drug during the course of the study.
* The subj is, in the opinion of the Institutional Principal Investigator, not an appropriate candidate for study participation.
* The subj participated in the study previously and was withdrawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2006-02-23 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay O. Boyle, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- India (2):
  - Amrita Institute of Sciences (AIMS), Kochi
  - Regional Cancer Center (RCC), Trivandrum

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: sulindac
  sulindac: Sulindac 150 mg po bid x 24 weeks
- Cohort 2: placebo
  Placebo: Placebo bid x 24 weeks
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 30 | 33
Completed | 30 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Continuous [Mean (Full Range); unit: years] | 54.5 [32 to 84] | 58.6 [28 to 84] | 56.6 [28 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 25 | 23 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 33 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 20 | 23 | 43
  Native Hawaiian or Other Pacific Islander | 7 | 8 | 15
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6
  India | 27 | 30 | 57

OUTCOME MEASURES:

1. Primary Outcome: - To Evaluate the Efficacy of Sulindac in Subjects With Early or Advanced Oral Premalignant Lesion (OPL) by Both Clinical Response (Reduction in Size of All Lesions) and Histological Response (Change in Histological Grade).
Time Frame: after 24 weeks of study drug
Population: Data were not collected
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Evaluate the Effect of Sulindac in Modulating the Expression of the Intermediate Biomarkers Ki67, p53 Proteins and DNA Ploidy After 24 Weeks of Treatment of Study Drug, and Again After 8 Weeks Off Study Drug.
Time Frame: after 24 weeks of study drug
Population: Data were not collected
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: To Evaluate the Correlation Between Baseline COX-2 Expression or DNA Ploidy With Clinical Response or Biomarker Modulation
Time Frame: baseline and after 24 weeks
Population: Data were not collected
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: To Evaluate the Safety of Chronic Dosing of Sulindac in This Subject Population
Time Frame: week 4, 8, 12, 16, 20 and 24
Population: Data were not collected
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: To Explore the Relationship Between Genetic Polymorphisms of Genes Involved in Carcinogenesis and Clinical or Biomarker Response to Sulindac
Time Frame: after 24 weeks
Population: Data were not collected
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 1/30 | 4/33
Serious Adverse Events (participants affected / at risk) | 2/30 | 4/33
Other Adverse Events (participants affected / at risk) | 13/30 | 13/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=30) | Cohort 2 (N=33)
Gastrointestinal, other (Gastrointestinal disorders) | 1 | 3
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 1 | 0
Death not assoc w CTCAE term- Death NOS (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=30) | Cohort 2 (N=33)
Constipation (Gastrointestinal disorders) | 1 | 1
Dermatology/Skin, other (Skin and subcutaneous tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Endocrine, other (Endocrine disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Gastritis (incl bile reflux gastritis) (Gastrointestinal disorders) | 0 | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 | 1
Hemorrhage/Bleeding, other (Injury, poisoning and procedural complications) | 0 | 2
Inf norm ANC/gr1/2 neut-Bronchitis NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Inf norm ANC/gr1/2 neut-Gingivitis(oral-gums) (Gastrointestinal disorders) | 1 | 0
Lymphatics - Other (specify) (Immune system disorders) | 0 | 1
Mucositis (Clin exam)- Oral cavity (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Ocular/Visual - Other (specify) (Eye disorders) | 1 | 0
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 | 0
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain - Head/headache (Nervous system disorders) | 1 | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain - Oral cavity (Gastrointestinal disorders) | 0 | 1
Pain - Other (specify) (General disorders) | 2 | 0
Pulm/upp respiratory - Other (spec) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT00299195/Prot_SAP_000.pdf